CLINICAL TRIAL: NCT00734162
Title: A Randomized, Double-Blind Evaluation of the Antiviral Efficacy, Safety, and Tolerability of Tenofovir Disoproxil Fumarate Versus Placebo in Adolescents With Chronic Hepatitis B Infection
Brief Title: Evaluation of Tenofovir Disoproxil Fumarate in Adolescents With Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-174-0115
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis B Virus (HBV)
Keywords: tenofovir; adolescents; chronic hepatitis B
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir disoproxil fumarate (TDF) (Experimental)
  Interventions: Drug: Tenofovir disoproxil fumarate (TDF)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate (TDF) — TDF administered as a 300-mg tablet once daily
  Other Names: Viread®
  Arms: Tenofovir disoproxil fumarate (TDF)
Drug: Placebo — TDF placebo tablet once daily
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the effectiveness, safety, and tolerability of tenofovir disoproxil fumarate (TDF) in adolescents (aged 12-17 years) with chronic hepatitis B virus (HBV) infection.

The optimal treatment for adolescents with chronic HBV infection is currently unknown. Treatment with interferon alfa, lamivudine, and adefovir dipivoxil in pediatric populations has been shown to be less than optimal. Further, the safety and efficacy of entecavir and telbivudine have not been established in patients < 16 years of age. A study evaluating TDF in adolescents (ages 12-17) was needed to assess the safety and efficacy of this agent in the treatment of chronic hepatitis B in this patient population. In addition, the study will help to further elucidate the pharmacokinetic (PK) and resistance profiles of TDF. Through their participation, study participants will help generate critical new information to help guide the most optimal treatment of chronic HBV infection in adolescents.

This is a randomized, double-blind study to evaluate the antiviral efficacy, safety, and tolerability of TDF versus placebo in adolescents with chronic HBV infection. TDF treatment-naive participants were randomized in a 1:1 ratio to TDF or placebo. After 72 weeks of blinded treatment, participants were to switch to open-label TDF for an additional 2.5 years of treatment, provided that no safety concerns are identified by the Independent Data Monitoring Committee monitoring the study.

ELIGIBILITY:
Inclusion Criteria

* Male or female, 12 through 17 years of age, inclusive (consent of parent/legal guardian required)
* Documented chronic HBV infection
* HBeAg positive or HBeAg negative
* Weight > 35 kg
* Able to swallow oral tablets
* HBV DNA > 100,000 copies/mL (polymerase chain reaction (PCR) method)
* Alanine aminotransferase (ALT) > 2 × upper limit of normal (ULN) at screening, OR any history of ALT > 2 × ULN over the past 24 months
* Willing and able to provide written informed consent/assent (child and parent/legal guardian)
* Negative serum pregnancy test (for postmenarchal females only)
* Estimated glomerular filtration rate (creatinine clearance [using the Schwartz formula]) > 80 mL/min/1.73m^2
* Adequate hematologic function (absolute neutrophil count ≥ 1,500/mm^3; hemoglobin ≥ 10.0 g/dL)
* No prior TDF therapy (participants may have received prior interferon or oral anti-HBV nucleoside/nucleotide therapy; participants must have discontinued interferon therapy ≥ 6 months prior to screening; participants experienced on anti-HBV nucleoside/nucleotide therapy must have discontinued therapy ≥ 16 weeks prior to screening to avoid flare if randomized to the placebo arm)

Exclusion Criteria

* Pregnant women, women who are breast feeding or who believe they may wish to become pregnant during the course of the study
* Males and females of reproductive potential who are not willing to use an effective method of contraception during the study
* Decompensated liver disease
* Receipt of interferon (pegylated or not) therapy within 6 months of the Screening Visit
* Receipt of anti-HBV nucleoside/nucleotide therapy within 16 weeks of the Screening Visit
* Alpha fetoprotein > 50 ng/mL
* Evidence of hepatocellular carcinoma (HCC)
* Coinfection with HIV, hepatitis C virus (HCV), or hepatitis D virus (HDV)
* History of significant renal disease (eg, nephrotic syndrome, renal dysgenesis, polycystic kidney disease, congenital nephrosis, acute tubular necrosis, other renal disease)
* History of significant bone disease (eg, osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, osteochondroses, multiple bone fractures)
* Significant cardiovascular, pulmonary, or neurological disease
* Evidence of a gastrointestinal malabsorption syndrome that may interfere with absorption of orally administered medications
* History of solid organ or bone marrow transplantation
* Ongoing therapy with nephrotoxic agents, competitors of renal excretion, systemic chemotherapeutic agents, systemic corticosteroids, interleukin-2 (IL-2), or other immunomodulating or investigational agents
* Known hypersensitivity to the study drugs, the metabolites or formulation excipients
* Any other condition (including alcohol or substance abuse) or prior therapy that, in the opinion of the Investigator, would make the participants unsuitable for the study or unable to comply with dosing requirements

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benedetta Massetto, MD, PhD, Study Director — Gilead Sciences
Locations (21):
- United States (3):
  - Children's Hospital & Research Center at Oakland, Oakland, California
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital & Regional Medical Center, d/b/a Seattle Children's Research Institute, Seattle, Washington
- Bulgaria (2):
  - Multiprofile Hospital for Active Treatment Sveti Georgi, Plovdiv
  - Clinic of Gastroenterology, Specialized Hospital for Active Treatment of Pediatric Diseases, Sofia, Sofia
- France (2):
  - Hopital Femmes Meres Enfants, Bron
  - Hôpital Claude Huriez, Lille
- Poland (8):
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny Akademii Medycznej w Bialymstoku, Bialystok
  - Wojewodzki Specjalistyczny Szpital im Bieganskiego, Bydgoszcz
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. T. Browicza, Bydgoszcz
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Samodzielny Publiczny Szpital Kliniczny im. Karola Johschera, Poznan
  - Specjalistyczny Zespol Opieki Zdrowotnej nad Matka i Dzieckiem, Poznan
  - Wojewodzki Szpital Zakazny, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Wroclaw
- Romania (3):
  - Fundeni Clinical Institute, Bucharest
  - Institute for Infectious Diseases, Bucharest
  - Cluj Childrens Emergency Hospital, Napaco
- Spain (2):
  - Hosp Univ y Politecnico La Fe de Valencia, Madrid
  - Hospital Universitario De Getafe, Madrid
- Ege Universitesi Tip Fakultesi Hastanesi, Izmir, Turkey (Türkiye)

REFERENCES:
- [Result] Murray KF, Szenborn L, Wysocki J, Rossi S, Corsa AC, Dinh P, McHutchison J, Pang PS, Luminos LM, Pawlowska M, Mizerski J. Randomized, placebo-controlled trial of tenofovir disoproxil fumarate in adolescents with chronic hepatitis B. Hepatology. 2012 Dec;56(6):2018-26. doi: 10.1002/hep.25818. Epub 2012 Aug 27. PMID 22544804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 3 sites in the United States, 8 sites in Poland, 3 sites in Romania, 2 sites in Bulgaria, 2 sites in France, 2 sites in Spain, and 1 site in Turkey. The first participant was screened on 03 December 2008. The last study visit occurred on 02 December 2015.
Pre-assignment Details: 149 participants were screened.
Groups:
- TDF 12-14 Years: Tenofovir disoproxil fumarate (TDF) 300 mg tablet once daily in participants 12-14 years of age in the Randomized Phase, followed by TDF 300 mg tablet once daily in the Open-Label Phase
- TDF 15-17 Years: TDF 300 mg tablet once daily in participants 15-17 years of age in the Randomized Phase, followed by TDF 300 mg tablet once daily in the Open-Label Phase
- Placebo 12-14 Years: TDF placebo tablet once daily in participants 12-14 years of age in the Randomized Phase, followed by TDF 300 mg tablet once daily in the Open-Label Phase
- Placebo 15-17 Years: TDF placebo tablet once daily in participants 15-17 years of age in the Randomized Phase, followed by TDF 300 mg tablet once daily in the Open-Label Phase
Period: Randomized Phase (Through Week 72)
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years
Started | 10 | 42 | 13 | 41
Completed | 10 | 41 | 13 | 37
Not Completed | 0 | 1 | 0 | 4
Not completed — Investigator's Discretion | 0 | 1 | 0 | 2
Not completed — Per protocol ALT elevation | 0 | 0 | 0 | 2
Period: Open-Label Phase
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years
Started | 10 | 41 | 13 | 39 (2 participants switched to open-label treatment before completing double-blind period (elevated ALT))
Completed | 7 | 39 | 12 | 36
Not Completed | 3 | 2 | 1 | 3
Not completed — Safety, Tolerability or Efficacy Reasons | 1 | 0 | 0 | 0
Not completed — Withdrew Consent | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0 | 1
Not completed — Did Not Meet Entrance Criteria | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TDF 12-14 Years: TDF 300 mg tablet once daily in participants 12-14 years of age in the Randomized Phase, followed by TDF 300 mg tablet once daily in the Open-Label Phase
- Total: Total of all reporting groups
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (0.82) | 16.1 (0.75) | 13.2 (0.69) | 15.9 (0.82) | 15.4 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 4 | 15 | 33
  Male | 7 | 31 | 9 | 26 | 73
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1 | 0 | 2
  Black | 0 | 1 | 0 | 0 | 1
  White | 10 | 39 | 12 | 37 | 98
  Other | 0 | 1 | 0 | 4 | 5
Region of Enrollment [Number; unit: participants]
  Bulgaria | 0 | 3 | 3 | 1 | 7
  France | 0 | 1 | 0 | 1 | 2
  Poland | 6 | 31 | 6 | 31 | 74
  Romania | 4 | 4 | 2 | 4 | 14
  Spain | 0 | 0 | 0 | 2 | 2
  Turkey | 0 | 1 | 1 | 0 | 2
  United States | 0 | 2 | 1 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Europe | 10 | 40 | 12 | 39 | 101
  North America | 0 | 2 | 1 | 2 | 5
Alanine aminotransferase (ALT) level at baseline [Mean (Standard Deviation); unit: U/L] | 77 (54.8) | 106 (116.4) | 101 (95.4) | 101 (89.5) | 101 (98.5)
ALT normal at baseline [Number; unit: participants] — The upper limit of normal (ULN) was 43 U/L for males and 34 U/L for females.
  participants
    Normal | 3 | 14 | 4 | 8 | 29
    Abnormal | 7 | 28 | 9 | 33 | 77
HBV Genotype [Number; unit: participants]
  Genotype A | 5 | 30 | 5 | 29 | 69
  Genotype B | 0 | 1 | 1 | 1 | 3
  Genotype C | 0 | 1 | 0 | 0 | 1
  Genotype D | 5 | 10 | 7 | 11 | 33
Hepatitis B e Antigen (HBeAg) status at baseline [Number; unit: participants]
  Negative | 1 | 3 | 0 | 6 | 10
  Positive | 9 | 39 | 13 | 35 | 96
HBV DNA level at baseline [Mean (Standard Deviation); unit: Log_10 copies/mL] | 8.26 (1.455) | 7.95 (1.421) | 8.61 (1.166) | 8.12 (1.451) | 8.13 (1.403)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL at Week 72
Description: The percentage of participants with HBV DNA < 400 copies/mL at Week 72 was summarized by treatment and age group (grouped by baseline age for analysis), using the missing = failure (M = F) analysis with the double-blind efficacy evaluation (DBEE) algorithm.
  In the M = F analysis method, all missing data were considered as failure to meet the outcome measure threshold. This method was combined with the DBEE algorithm, which included all available data for the double-blind period, and any data for the open-label period were not included; data generated during treatment-free follow-up from subjects who achieved HBsAg loss and entered treatment-free follow-up during double-blind treatment period were included.
Time Frame: Week 72
Population: Full Analysis Set: participants who were randomized and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- Total TDF 12-17 Years: TDF 300 mg tablet once daily in participants 12-17 years of age in the Randomized Phase, followed by TDF 300 mg tablet once daily in the Open-Label Phase
- Total Placebo 12-17 Years: TDF placebo tablet once daily in participants 12-17 years of age in the Randomized Phase, followed by TDF 300 mg tablet once daily in the Open-Label Phase
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 52 | 54
percentage of participants | 90.0 | 88.1 | 0 | 0 | 88.5 | 0
Statistical Analysis 1: Comparison: TDF 12-14 Years vs TDF 15-17 Years vs Placebo 12-14 Years vs Placebo 15-17 Years; Analysis is the difference between treatment groups in the proportion of participants who met the outcome measure criterion, controlling for randomization age group; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — A p-value of < 0.05 was considered statistically significant

2. Primary Outcome: Percentage of Participants With at Least a 6% Decrease From Baseline in Bone Mineral Density (BMD) of the Spine at Week 72
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
  In contrast with what was previously reported in the interim results posting, 1 participant met the primary safety endpoint of at least a 6% decrease from baseline in spine BMD at Week 72, based on the final BMD data analysis. The apparent discrepancy was due to the correction factor applied to the subject-specific BMD calculations performed at the time of the Interim Week 72 clinical study report that could not take into account the actual Week 72 phantom data (ie, calibration test used in longitudinal clinical trials to monitor and adjust for shifts in the dual-energy x-ray absorptiometry (DXA) scanner calibration over time), which were not provided by the site at that time. The correction factor applied to the final analysis has been properly based on all phantom data through the end of Week 72, as well as through the end of Week 192.
Time Frame: Baseline to Week 72
Population: Safety Analysis Set: participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 52 | 54
percentage of participants | 0 | 2.4 | 0 | 0 | 1.9 | 0

3. Secondary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL at Weeks 48, 96, 144, and 192
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis) using the missing = failure method.
Time Frame: Weeks 48, 96, 144, and 192
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 52 | 54
percentage of participants
  Week 48 | 90.0 | 85.7 | 0 | 0 | 86.5 | 0
  Week 96 | 90.0 | 88.1 | 53.8 | 68.3 | 88.5 | 64.8
  Week 144 | 100.0 | 90.5 | 69.2 | 85.4 | 92.3 | 81.5
  Week 192 | 90.0 | 85.7 | 76.9 | 73.2 | 86.5 | 74.1

4. Secondary Outcome: Percentage of Participants With Normal Alanine Aminotransferase (ALT) at Weeks 48, 72, 96, 144, and 192
Description: as for outcome 3
Time Frame: Weeks 48, 72, 96, 144, and 192
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 52 | 54
percentage of participants
  Week 48 | 70.0 | 76.2 | 30.8 | 26.8 | 75.0 | 27.8
  Week 72 | 80.0 | 76.2 | 30.8 | 41.5 | 76.9 | 38.9
  Week 96 | 80.0 | 76.2 | 69.2 | 65.9 | 76.9 | 66.7
  Week 144 | 60.0 | 71.4 | 69.2 | 75.6 | 69.2 | 74.1
  Week 192 | 80.0 | 71.4 | 84.6 | 75.6 | 73.1 | 77.8

5. Secondary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL and Normal ALT at Weeks 48, 72, 96, 144, and 192
Description: as for outcome 3
Time Frame: Weeks 48, 72, 96, 144, and 192
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 52 | 54
percentage of participants
  Week 48 | 70.0 | 69.0 | 0 | 0 | 69.2 | 0
  Week 72 | 80.0 | 69.0 | 0 | 0 | 71.2 | 0
  Week 96 | 80.0 | 73.8 | 46.2 | 51.2 | 75.0 | 50.0
  Week 144 | 60.0 | 69.0 | 53.8 | 68.3 | 67.3 | 64.8
  Week 192 | 80.0 | 64.3 | 69.2 | 63.4 | 67.3 | 64.8

6. Secondary Outcome: Percentage of Participants With HBV DNA < 169 Copies/mL at Weeks 48, 72, 96, 144, and 192
Description: as for outcome 3
Time Frame: Weeks 48, 72, 96, 144, and 192
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 52 | 54
percentage of participants
  Week 48 | 80.0 | 81.0 | 0 | 0 | 80.8 | 0
  Week 72 | 90.0 | 83.3 | 0 | 0 | 84.6 | 0
  Week 96 | 90.0 | 88.1 | 53.8 | 63.4 | 88.5 | 61.1
  Week 144 | 90.0 | 88.1 | 69.2 | 82.9 | 88.5 | 79.6
  Week 192 | 90.0 | 83.3 | 76.9 | 73.2 | 84.6 | 74.1

7. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Weeks 48, 72, 96, 144, and 192
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis), using the M = F.
Time Frame: Baseline; Weeks 48, 72, 96, 144, and 192
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 52 | 54
percentage of participants
  Week 48 | 0 | 0 | 0 | 0 | 0 | 0
  Week 72 | 0 | 2.4 | 0 | 0 | 1.9 | 0
  Week 96 | 0 | 2.4 | 0 | 0 | 1.9 | 0
  Week 144 | 0 | 2.4 | 0 | 0 | 1.9 | 0
  Week 192 | 0 | 2.4 | 0 | 0 | 1.9 | 0

8. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Weeks 48, 72, 96, 144, and 192
Description: HBsAg seroconversion was defined as change of detectable antibody to HBsAg from negative to positive. Data were summarized by treatment and age group (grouped by baseline age for analysis), using the M = F.
Time Frame: Baseline; Weeks 48, 72, 96, 144, and 192
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 52 | 54
percentage of participants
  Week 48 | 0 | 0 | 0 | 0 | 0 | 0
  Week 72 | 0 | 2.4 | 0 | 0 | 1.9 | 0
  Week 96 | 0 | 2.4 | 0 | 0 | 1.9 | 0
  Week 144 | 0 | 2.4 | 0 | 0 | 1.9 | 0
  Week 192 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants With at Least a 6% Decrease From Baseline in Spine BMD at Weeks 48, 96, 144, and 192
Description: The percentage of participants reported is the cumulative incidence from baseline to the respective time point. Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Weeks 48, 96, 144, and 192
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 52 | 54
percentage of participants
  Week 48 | 0 | 0 | 0 | 0 | 0 | 0
  Week 96 | 0 | 2.4 | 0 | 0 | 1.9 | 0
  Week 144 | 0 | 2.4 | 0 | 0 | 1.9 | 0
  Week 192 | 0 | 4.8 | 0 | 4.9 | 3.8 | 3.7

10. Secondary Outcome: Percentage of Participants With at Least a 6% Decrease From Baseline in Whole Body BMD at Weeks 48, 72, 96, 144, and 192
Description: as for outcome 9
Time Frame: Baseline; Weeks 48, 72, 96, 144, and 192
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 42 | 13 | 41 | 52 | 54
percentage of participants
  Week 48 | 0 | 0 | 0 | 0 | 0 | 0
  Week 72 | 0 | 0 | 0 | 0 | 0 | 0
  Week 96 | 0 | 0 | 0 | 0 | 0 | 0
  Week 144 | 0 | 0 | 0 | 2.4 | 0 | 1.9
  Week 192 | 0 | 0 | 0 | 2.4 | 0 | 1.9

11. Secondary Outcome: Percent Change From Baseline in Spine Bone Mineral Density (BMD) at Week 48
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 41 | 12 | 37 | 51 | 49
percentage change | 9.234 (3.4782) | 2.114 (3.6023) | 9.038 (6.6575) | 4.435 (4.9091) | 3.510 (4.5507) | 5.562 (5.6772)

12. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 72
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 72
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 41 | 12 | 37 | 51 | 49
percentage change | 11.516 (3.8818) | 3.589 (4.5633) | 14.131 (9.9563) | 6.117 (6.0624) | 5.144 (5.4291) | 8.080 (7.8996)

13. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 96
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 40 | 11 | 39 | 50 | 50
percentage change | 13.811 (4.6712) | 4.196 (4.8021) | 16.687 (10.4359) | 4.272 (7.0463) | 6.119 (6.1200) | 7.003 (9.3658)

14. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 144
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 144
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 39 | 10 | 38 | 49 | 48
percentage change | 19.224 (8.7594) | 5.289 (5.8084) | 21.346 (13.4709) | 6.144 (8.3286) | 8.133 (8.5611) | 9.311 (11.3262)

15. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 192
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 192
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 37 | 11 | 35 | 46 | 46
percentage change | 23.933 (8.5166) | 6.673 (7.2870) | 25.036 (14.2346) | 6.867 (9.3736) | 10.050 (10.1637) | 11.212 (13.1459)

16. Secondary Outcome: Percent Change From Baseline in Whole Body BMD at Week 48
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 39 | 13 | 37 | 48 | 50
percentage change | 5.123 (3.8309) | 1.339 (1.9324) | 5.470 (3.4958) | 3.236 (2.8573) | 2.048 (2.7830) | 3.817 (3.1576)

17. Secondary Outcome: Percent Change From Baseline in Whole Body BMD at Week 72
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 72
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 41 | 13 | 38 | 50 | 51
percentage change | 7.282 (3.9156) | 2.141 (2.6284) | 8.480 (4.4770) | 4.335 (3.4073) | 3.067 (3.4819) | 5.391 (4.0902)

18. Secondary Outcome: Percent Change From Baseline in Whole Body BMD at Week 96
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 40 | 12 | 38 | 49 | 50
percentage change | 8.034 (3.4973) | 3.023 (3.2063) | 10.056 (5.4296) | 4.291 (4.3195) | 3.943 (3.7730) | 5.675 (5.1858)

19. Secondary Outcome: Percent Change From Baseline in Whole Body BMD at Week 144
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 144
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 38 | 11 | 38 | 47 | 49
percentage change | 10.940 (4.8819) | 3.529 (3.1734) | 12.638 (5.9973) | 4.730 (5.2213) | 4.949 (4.5753) | 6.505 (6.2944)

20. Secondary Outcome: Percent Change From Baseline in Whole Body BMD at Week 192
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 192
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 8 | 35 | 12 | 34 | 43 | 46
percentage change | 13.923 (4.6139) | 4.295 (3.7318) | 14.797 (6.4993) | 4.549 (5.4494) | 6.086 (5.4029) | 7.223 (7.2666)

21. Secondary Outcome: Change From Baseline in Z-score for Spine BMD at Week 48
Description: To assess any effect of treatment on growth, Z-scores were used to express the deviation from a reference population for lumbar spine BMD. A Z-score of 0 indicated that a subject was typical of the population for their age, ethnicity, and gender. A negative Z-score indicated that the subject's recorded value was lower than typical for their age, ethnicity, and gender. A positive Z-score indicates that the subject's recorded value was higher than typical for their age, ethnicity, and gender. Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 41 | 12 | 37 | 51 | 49
z-score | 0.02 (0.247) | -0.10 (0.255) | 0.04 (0.393) | 0.05 (0.322) | -0.08 (0.256) | 0.05 (0.337)

22. Secondary Outcome: Change From Baseline in Z-score for Spine BMD at Week 72
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 72
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 41 | 12 | 37 | 51 | 49
z-score | -0.10 (0.312) | -0.05 (0.325) | 0.09 (0.498) | 0.10 (0.339) | -0.06 (0.320) | 0.10 (0.378)

23. Secondary Outcome: Change From Baseline in Z-score for Spine BMD at Week 96
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 40 | 11 | 39 | 50 | 50
z-score | -0.19 (0.365) | -0.07 (0.356) | -0.02 (0.498) | -0.13 (0.414) | -0.10 (0.357) | -0.11 (0.431)

24. Secondary Outcome: Change From Baseline in Z-score for Spine BMD at Week 144
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 144
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 10 | 39 | 10 | 38 | 49 | 48
z-score | -0.20 (0.560) | -0.05 (0.417) | -0.16 (0.625) | -0.04 (0.405) | -0.08 (0.447) | -0.06 (0.455)

25. Secondary Outcome: Change From Baseline in Z-score for Spine BMD at Week 192
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 192
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 37 | 11 | 35 | 46 | 46
z-score | -0.24 (0.518) | 0.08 (0.544) | -0.26 (0.654) | -0.05 (0.504) | 0.02 (0.548) | -0.10 (0.543)

26. Secondary Outcome: Change From Baseline in Z-score for Whole Body BMD at Week 48
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 39 | 13 | 37 | 48 | 50
z-score | 0.02 (0.426) | -0.15 (0.257) | 0.10 (0.370) | 0.04 (0.308) | -0.12 (0.298) | 0.05 (0.322)

27. Secondary Outcome: Change From Baseline in Z-score for Whole Body BMD at Week 72
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 72
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 41 | 13 | 38 | 50 | 51
z-score | 0.02 (0.398) | -0.19 (0.338) | 0.20 (0.450) | 0.06 (0.306) | -0.16 (0.355) | 0.09 (0.349)

28. Secondary Outcome: Change From Baseline in Z-score for Whole Body BMD at Week 96
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 40 | 12 | 38 | 49 | 50
z-score | -0.12 (0.294) | -0.19 (0.451) | 0.09 (0.528) | -0.06 (0.432) | -0.18 (0.424) | -0.03 (0.456)

29. Secondary Outcome: Change From Baseline in Z-score for Whole Body BMD at Week 144
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 144
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 38 | 11 | 38 | 47 | 49
z-score | -0.27 (0.431) | -0.21 (0.473) | -0.06 (0.554) | -0.16 (0.468) | -0.22 (0.462) | -0.14 (0.484)

30. Secondary Outcome: Change From Baseline in Z-score for Whole Body BMD at Week 192
Description: Data were summarized by treatment and age group (grouped by baseline age for analysis).
Time Frame: Baseline; Week 192
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 8 | 35 | 12 | 34 | 43 | 46
z-score | -0.34 (0.499) | -0.11 (0.524) | -0.21 (0.486) | -0.19 (0.517) | -0.16 (0.521) | -0.19 (0.504)

31. Secondary Outcome: Number of Participants With Changes in Drug-Resistant Mutations During the Study
Description: The number of participants with changes in drug-resistant mutations during the study was summarized.
Time Frame: Baseline through Week 192
Population: Participants with HBV DNA ≥ 400 copies/mL, with confirmed virologic breakthrough (defined as 2 consecutive increases in HBV DNA of at least 10-fold from nadir, or confirmed values ≥ 400 copies/mL after being < 400 copies/mL while on study medication), or subjects who discontinued early (after Week 24 with HBV DNA ≥ 400 copies/mL) were analyzed.
Measure: Number; unit: participants
Arm/Group | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 52 | 54
participants
  New TDF Drug-Resistant Mutations | 0 | 0
  Enrichment of TDF Drug-Resistant Mutations | 0 | 0

32. Secondary Outcome: Percentage of Participants Who Were HBeAg-Positive at Baseline and Who Had HBeAg Loss at Weeks 48, 72, 96, 144, and 192
Description: as for outcome 3
Time Frame: Baseline; Weeks 48, 72, 96, 144, and 192
Population: Participants in the Full Analysis Set who were HBeAg-positive at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 39 | 13 | 35 | 48 | 48
percentage of participants
  Week 48 | 11.1 | 17.9 | 7.7 | 8.6 | 16.7 | 8.3
  Week 72 | 11.1 | 23.1 | 23.1 | 11.4 | 20.8 | 14.6
  Week 96 | 44.4 | 30.8 | 38.5 | 28.6 | 33.3 | 31.3
  Week 144 | 44.4 | 38.5 | 53.8 | 34.3 | 39.6 | 39.6
  Week 192 | 33.3 | 43.6 | 53.8 | 37.1 | 41.7 | 41.7

33. Secondary Outcome: Percentage of Participants Who Were HBeAg-Positive at Baseline and Who Had HBeAg Seroconversion at Weeks 48, 72, 96, 144, and 192
Description: as for outcome 3
Time Frame: Baseline; Weeks 48, 72, 96, 144, and 192
Population: Participants in the Full Analysis Set who were HBeAg-positive at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 39 | 13 | 35 | 48 | 48
percentage of participants
  Week 48 | 11.1 | 15.4 | 7.7 | 8.6 | 14.6 | 8.3
  Week 72 | 11.1 | 23.1 | 23.1 | 11.4 | 20.8 | 14.6
  Week 96 | 44.4 | 30.8 | 38.5 | 25.7 | 33.3 | 29.2
  Week 144 | 33.3 | 38.5 | 53.8 | 34.3 | 37.5 | 39.6
  Week 192 | 33.3 | 38.5 | 53.8 | 37.1 | 37.5 | 41.7

34. Secondary Outcome: Percentage of Participants Who Were HBeAg-Positive at Baseline Who Had HBV DNA < 400 Copies/mL, Normal ALT, and HBeAg Loss/Seroconversion at Weeks 48, 72, 96, 144, and 192
Description: as for outcome 3
Time Frame: Baseline; Weeks 48, 72, 96, 144, and 192
Population: Participants in the Full Analysis Set who were HBeAg-positive at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 9 | 39 | 13 | 35 | 48 | 48
percentage of participants
  Week 48 | 11.1 | 12.8 | 0 | 0 | 12.5 | 0
  Week 72 | 11.1 | 15.4 | 0 | 0 | 14.6 | 0
  Week 96 | 44.4 | 28.2 | 30.8 | 22.9 | 31.3 | 25.0
  Week 144 | 22.2 | 30.8 | 46.2 | 25.7 | 29.2 | 31.3
  Week 192 | 33.3 | 28.2 | 46.2 | 25.7 | 29.2 | 31.3

35. Secondary Outcome: Percentage of Participants With Abnormal ALT at Baseline Who Had Normalized ALT at Weeks 48, 72, 96, 144, and 192
Description: as for outcome 3
Time Frame: Baseline; Weeks 48, 72, 96, 144, and 192
Population: Participants in the Full Analysis Set with abnormal ALT at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 7 | 28 | 9 | 33 | 35 | 42
percentage of participants
  Week 48 | 85.7 | 71.4 | 11.1 | 21.2 | 74.3 | 19.0
  Week 72 | 85.7 | 71.4 | 22.2 | 33.3 | 74.3 | 31.0
  Week 96 | 85.7 | 78.6 | 66.7 | 63.6 | 80.0 | 64.3
  Week 144 | 57.1 | 71.4 | 66.7 | 72.7 | 68.6 | 71.4
  Week 192 | 85.7 | 75.0 | 77.8 | 69.7 | 77.1 | 71.4

36. Secondary Outcome: Percentage of Participants With Abnormal ALT at Baseline Who Had HBV DNA < 400 Copies/mL and Normalized ALT at Weeks 48, 72, 96, 144, and 192
Description: as for outcome 3
Time Frame: Baseline; Weeks 48, 72, 96, 144, and 192
Population: Participants in the Full Analysis Set with abnormal ALT at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 7 | 28 | 9 | 33 | 35 | 42
percentage of participants
  Week 48 | 85.7 | 71.4 | 0 | 0 | 74.3 | 0
  Week 72 | 85.7 | 71.4 | 0 | 0 | 74.3 | 0
  Week 96 | 85.7 | 78.6 | 55.6 | 54.5 | 80.0 | 54.8
  Week 144 | 57.1 | 71.4 | 66.7 | 69.7 | 68.6 | 69.0
  Week 192 | 85.7 | 67.9 | 77.8 | 57.6 | 71.4 | 61.9

37. Secondary Outcome: Percentage of Participants Who Were HBeAg-Positive With Abnormal ALT at Baseline Who Had HBV DNA < 400 Copies/mL, Normalized ALT, and HBeAg Loss/Seroconversion at Weeks 48, 72, 96, 144, and 192
Description: as for outcome 3
Time Frame: Baseline; Weeks 48, 72, 96, 144, and 192
Population: Participants in the Full Analysis Set who were HBeAg-Positive with abnormal ALT at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 12-14 Years | TDF 15-17 Years | Placebo 12-14 Years | Placebo 15-17 Years | Total TDF 12-17 Years | Total Placebo 12-17 Years
Number analyzed (Participants) | 6 | 27 | 9 | 33 | 33 | 42
percentage of participants
  Week 48 | 16.7 | 18.5 | 0 | 0 | 18.2 | 0
  Week 72 | 16.7 | 22.2 | 0 | 0 | 21.2 | 0
  Week 96 | 50.0 | 33.3 | 33.3 | 24.2 | 36.4 | 26.2
  Week 144 | 33.3 | 29.6 | 55.6 | 27.3 | 30.3 | 33.3
  Week 192 | 50.0 | 29.6 | 55.6 | 27.3 | 33.3 | 33.3

ADVERSE EVENTS:
Time Frame: Baseline through end of the Open-Label Phase (up to 4 years)
Description: Safety Analysis Set
Groups:
- Double-Blind TDF: Adverse events reported in this group occurred during the Randomized Phase (+7 days for participants who did not continue to the Open-Label Phase) and includes all participants who received double-blind TDF during the Randomized Phase of the study.
- Double-Blind Placebo: Adverse events reported in this group occurred during the Randomized Phase (+7 days for participants who did not continue to the Open-Label Phase) and includes all participants who received placebo during the Randomized Phase of the study.
- Open-Label TDF-TDF: Adverse events reported in this group occurred during the Open-Label Phase and includes all participants who received double-blind TDF during the Randomized Phase of the study and continued to the Open-Label Phase.
- Open-Label Placebo-TDF: Adverse events reported in this group occurred during the Open-Label Phase and includes all participants who received placebo during the Randomized Phase of the study and continued to the Open-Label Phase.
Arm/Group | Double-Blind TDF | Double-Blind Placebo | Open-Label TDF-TDF | Open-Label Placebo-TDF
Serious Adverse Events (participants affected / at risk) | 5/52 | 11/54 | 8/51 | 10/52
Other Adverse Events (participants affected / at risk) | 34/52 | 40/54 | 30/51 | 31/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind TDF (N=52) | Double-Blind Placebo (N=54) | Open-Label TDF-TDF (N=51) | Open-Label Placebo-TDF (N=52)
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 7 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase abnormal (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Glucose urine present (Investigations) | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Drug dependence (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind TDF (N=52) | Double-Blind Placebo (N=54) | Open-Label TDF-TDF (N=51) | Open-Label Placebo-TDF (N=52)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 5 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 7 | 1 | 9
Constipation (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 3 | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 3 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 1 | 2
Bronchitis (Infections and infestations) | 2 | 1 | 6 | 4
Gastroenteritis (Infections and infestations) | 2 | 2 | 0 | 5
Herpes zoster (Infections and infestations) | 0 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 12 | 6 | 12
Pharyngitis (Infections and infestations) | 15 | 11 | 9 | 13
Respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 3
Rhinitis (Infections and infestations) | 5 | 3 | 3 | 1
Tonsillitis (Infections and infestations) | 2 | 4 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 7 | 3 | 7
Viral infection (Infections and infestations) | 0 | 0 | 4 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 5 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 0 | 2 | 1
Headache (Nervous system disorders) | 2 | 9 | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 4 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 10 | 2 | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years